CLINICAL TRIAL: NCT06283862
Title: MIVetsCan: Cannabis Coaching for Veteran Pain Management Trial (Phase 2)
Brief Title: MIVetsCan: Can-Coach Trial (Phase 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan, State of, Licensing and Regulatory Affairs (Unknown)
Responsible Party: Principal Investigator, Kevin Boehnke, Research Assistant Professor, Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00231159b; VMR2022-03 (Other Grant/Funding Number: Michigan, State of, Licensing and Regulatory Affairs, Department of 573000)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Veteran; Cannabis; Cannabidiol
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to immediately receive 4 sessions of tailored guidance or to receive it after 12 weeks, as a waitlist control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Education (Experimental): Education sessions starting ~ week 4 of trial
  Interventions: Behavioral: Educational Session
- Waitlist Control - delayed education (Other): Education sessions starting ~ week 12 of trial
  Interventions: Behavioral: Educational Session

INTERVENTIONS:
Behavioral: Educational Session — The initial session will last about 45 to 60 minutes. The subsequent 3 sessions are anticipated to take about 20-30 minutes.

SUMMARY:
The goal of the MIVetsCan Can-Coach Trial is to test four coaching sessions to help Veterans with chronic pain use their own cannabis products more effectively to manage pain and related symptoms.

DETAILED DESCRIPTION:
All study interactions will be done virtually.

ELIGIBILITY:
Inclusion Criteria:

* United States Veteran
* Experiencing chronic pain (pain lasting 3 or more months)
* Moderate to severe chronic pain
* Are planning or currently using cannabidiol (CBD) or cannabis products for pain management
* Able to read and speak English sufficiently to allow for informed consent and active participation in the educational intervention sessions
* Willingness to attend all study visits (conducted virtually)
* Willingness to fill out periodic assessments via smartphone to assess symptom status and cannabis use (protocol has more details)

Exclusion Criteria:

* Inability to provide informed consent (e.g., cognitive impairment, unable to sufficiently communicate in English)
* Participant states participant is pregnant
* Current diagnosis or past history of a psychotic disorder (schizophrenia spectrum, except substance/medication -induced or due to another condition)
* Current diagnosis or past history of bipolar disorder
* Unable to attend study visits
* Risk for imminent harm - Suicidal ideation or wish to die as assessed with the Positive and Negative Suicide Ideation (PANSI) questionnaire and further risk assessment by study team members
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) score | Up to 14 weeks

SECONDARY OUTCOMES:
Self-report of pain (intensity or severity) from a numerical rating scale of 0-10 | Up to 14 weeks
  Self report of pain from a numerical rating scale of 0-10 over 7 day epochs where a higher number score indicates more pain
Anxiety as measured by the score on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile version 2.1 | Up to 14 weeks
Pain interference trends as measured by the score on the PROMIS-29 Profile version 2.1 | Up to 14 weeks
Sleep disturbance as measured by the score on the PROMIS-29 Profile version 2.1 | Up to 14 weeks
Suicidal ideation as measured by the Positive and Negative Suicide Ideation (PANSI) - Positive ideation | Up to 14 weeks
Suicidal ideation as measured by the Positive and Negative Suicide Ideation (PANSI) - Negative ideation | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Boehnke, PhD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No